CLINICAL TRIAL: NCT03591978
Title: Isolation of Circulating Pulmonary Cells in COPD and Its Relationship With Clinical Relevant Outcomes.
Brief Title: Isolation of Circulating Pulmonary Cells in COPD and Its Relationship With Clinical Relevant Outcomes (IbICEnCa)
Acronym: IbICEnCa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital de Alta Resolucion de Loja. Agencia Sanitaria Hospital de Poniente (Other); Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Enrique Herrera Viedma, Vice-Rector for Research and Transfer, Universidad de Granada
Other Study IDs: CPCEST001
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: COPD; COPD Exacerbation; COPD, Severe Early-Onset
Keywords: Disease progression; Circulating Pulmonary Cells
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Disease, Chronic Obstructive, Severe Early-Onset; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy non smokers: Healthy subjects with no respiratory disease and never smokers
  Interventions: Diagnostic Test: Isolation of Circulating Pulmonary Cells in peripheral blood
- Healthy smokers: Healthy subjects without respiratory disease and at least a cumulative tobacco consumption history of <10 pack-years
  Interventions: Diagnostic Test: Isolation of Circulating Pulmonary Cells in peripheral blood
- COPD: COPD patients (diagnosed as recommended by GOLD 2017 strategy) former or current smokers with at least >10 pack-years
  Interventions: Diagnostic Test: Isolation of Circulating Pulmonary Cells in peripheral blood

INTERVENTIONS:
Diagnostic Test: Isolation of Circulating Pulmonary Cells in peripheral blood — Blood samples from healthy volunteers will be collected in EDTA tubes (Vacutainer, BD Bioscience). CPC will be isolated according to previous patented method (P201730724)

SUMMARY:
We have demonstrated for the very first time that it is possible to isolate CPCs (circulating pulmonary cells) in patients with COPD in a sample of 17 patients (with a recovery rate of nearly 40%) and none of 10 healthy, non- smokers controls with a patented method [provisional Spanish Patent Application (P201730724)], based on liquid biopsy methodology (Romero Palacios et at, submitted 2017), showing that patients with COPD and isolation of CPCs have a more severe disease (expressed as higher BODEx index) and a trend towards a higher rate of decline of lung function as well as an increased rate of exacerbations, suggesting that CPCs isolation could be of value as a diagnostic and prognostic tool identifying patients with more active diseases. However, due to the small sample, no definitive conclusions could be made. Moreover, as there were no healthy smokers included in this study, we couldn´t evaluate if CPCs could be isolated in this type of population.

The fact that CPCs could be isolated in a group of patients with COPD and its relationship with greater severity suggests that this could be a marker of progression of the disease and could detect those patients more likely to benefit from newer antiinflamatory therapies(17)

DETAILED DESCRIPTION:
1. HYPOTHESIS 1.1. MAIN HYPOTHESIS.

   * CPCs isolation is frequent in COPD patients and also (to a lower level) in smokers without COPD but is not possible in healthy non-smokers.
   * CPCs isolation is related to important clinical outcomes in COPD. 1.2. SECONDARY HYPOTHESIS.
   * CPCs isolation in COPD is related to a higher rate of decline of lung function, measured by changes in FEV1 during a 3 year period.
   * CPCs isolation in COPD is related to indirect measures of emphysema (DLCO and kCO).
   * Isolation of CPCs in COPD patients is related to a higher risk of exacerbations during follow- up.
   * Isolation of CPCs in COPD is related to a higher burden of symptoms, measured by standardized questionnaires as CAT (COPD Assessment Test) and mMRC (modified Medical Research Council Scale).
   * Isolation of CPCs in COPD is more frequent as disease progress to a more severe disease.
   * Isolation of CPCs in COPD is related to a higher extent of radiologic emphysema, measured by %LAA (percentage of low attenuation areas).
2. OUTCOMES. 2.1. PRIMARY OUTCOME 2.1.1. To evaluate the prevalence of CPCs isolation in peripheral blood from COPD patients, smoking and non-smoking healthy controls with a patented liquid-biopsy technique.

2.2. SECONDARY OUTCOMES 2.2.1. To establish if there are differences between CPCs isolation rates from COPD patients, smoking and non-smoking healthy controls 2.2.2. To evaluate the relationship between CPCs isolation and the degree of parenchymal destruction and empyshema expresed as DLCO and kCO.

2.2.3. To evaluate the relationship between CPCs isolation and emphysema degree expressed as CT scan measurements (% LAA).

2.2.4. To evaluate the relationship between historical FEV1decline and CPCs isolation in COPD patients.

2.2.5. To evaluate the relationship between prospective 1 year FEV1 decline and CPCs isolation in COPD patients.

2.2.6. To evaluate the impact of CPCs isolation on deterioriation of HRQoL in COPD using CAT scores at baseline and change from baseline during 1 year follow- up.

2.2.7. To evaluate the rate of moderate and severe exacerbations during 1-year follow up between COPD patients with and without CPCs isolation after adjustment for confounding variables 2.2.8. To evaluate the time to first moderate and severe exacerbation during 1-year follow up between COPD patients with and without CPCs isolation after adjustment for confounding variables.

2.2.9. To evaluate the rate of moderate and severe exacerbations during 1-year follow up between subjects with and without CPCs isolation after adjustment for confounding variables 2.2.10. To evaluate if there are differences in the rate of CPCs isolation between those patients with early onset COPD (defined as those with COPD before 60 years of age) and those with normal onset COPD (defined as those with COPD after 60 years of age).

2.2.11. To evaluate the time to first moderate and severe exacerbation during 1-year follow up between subjects with and without CPCs isolation after adjustment for confounding variables 2.2.12. To evaluate the impact of CPCs isolation on deterioriation of HRQoL in smoking subjects using CAT scores at baseline and change from baseline during 1 year follow- up.

2.2.13. To evaluate the relationship between prospective 1 year FEV1 decline and CPCs isolation in smoking and non-smoking controls. 3. MATERIAL AND METHODS 3.1. STUDY DESIGN This study is designed as an observational, longitudinal study, with one-year follow up- recruiting participants in a respiratory out patients office.

3.2. STUDY POPULATION. 3.2.1. Healthy non- smokers (n=20): adults aged more than 35 years-old, never smokers, without any significant respiratory disease.

3.2.2. Healthy smokers (n=30): adults aged ≥ 35 years- old, former or current smokers with an smoking history of at least 10 pack- years, with normal lung function (FEV1/FVC >0.70 and FEV1 and FVC > 80% predicted).

3.2.3. COPD patients (n=100): adults aged ≥ 35 years- old, former or current smokers with an smoking history of at least 10 pack- years, with a 2 year previous COPD diagnosis (FEV1/FVC postbronchodilatador < 0.7) and regular inhaled treatment.

3.3. INCLUSION & EXCLUSION CRITERIA: 3.3.1. Inclusion criteria 3.3.1.1. Adults of >35 years-old. 3.3.1.2. Patients who have given written informed consent 3.3.1.3. Absence of respiratory infection or COPD exacerbation in the 4 previous weeks to baseline visit.

3.3.2. Exclusion criteria 3.3.2.1. Other respiratory condition apart from COPD, such as previous diagnosis of bronchial asthma, obstructive sleep apnoea, idiopathic pulmonary fibrosis, pulmonary tuberculosis, alpha1 antitrypsin deficiency.

3.3.2.2. Current or previous cancer history (even if the patient has been diagnosed >5 years and there is no evidence of recurrence of disease).

3.3.2.3. Unwillingness to perform pulmonary function test or CT scan. 3.3.2.4. Participation in another investigational study or clinical trial. 3.4. STUDY VARIABLES. 3.4.1. Demograhic variables: demographic data on sex, age, anthropometric characteristics, ethnicity.

3.4.2. Toxic habits: tobacco consumption (expressed as pack-years), current or former smoker, alcohol abuse history, drug abuse history.

3.4.3. Medical history: previous and concomitant diseases, age since diagnosis, history of cardiovascular disease, history of metabolic syndrome, comorbidity indexes (Charlson index, COTE index).

3.4.4. Pharmacology treatment: current oral pharmacological treatments (dose, frequency and exposure history), current inhaled treatments (dose, frequency and exposure history) classified as LAMA monotherapy, LABA monotherapy, ICS/LABA FDC, ICS/LABA non-FDC, LAMA/LABA FDC, LAMA/LABA nonFDC, single triple therapy (ICS/LABA/LAMA FDC), splited triple therapy (ICS/LABA plus LAMA), iPDE4.

3.4.5. Non- pharmacological treatment: oxygen use (daily hours, time since first prescription, oxygen flow), non-invasive mechanical ventilation (daily use, time since first prescription), pulmonary rehabilitation.

3.4.6. COPD variables: age at diagnosis, COPD phenotype (frequent exacerbator, chronic bronchitis, emphysema- predominant, ACO), GOLD 2017 grade (A-B-C-D) severity of airflow limitation (based on FEV1% predicted), severity of disease based on multidimensional scores (BODE, BODEx indexes), lung function decline (from previous 2 years to end of one-year follow up, expressed as annualized rate of decline of FEV1 in mL/yr).

3.4.7. COPD Exacerbations: moderate exacerbations are defined as a change in respiratory symptoms that goes beyond the daily variation and needs systemic corticosteroids and/or antibiotic prescription. Severe exacerbations are defined as a change in respiratory symptoms that goes beyond the daily variation and needs hospital admission or ED for more than 24 hours.

3.4.8. Pulmonary function tests (PFTs):

* Spirometric measurements (FEV1 mL, FEV1% predicted, FVC mL, FVC% predicted, FEV1/FVC) and post bronchodilator (∆ FEV1mL; ∆ FEV1%) after inhalation of 400 mcgr of salbutamol.
* Body-plettismography measurements: FRC (expressed as mL and % predicted), RV (expressed as mL and % predicted), TLC (expressed as mL and % predicted) and RV/TLC ratio.
* Difussion capacity transfer for CO measurements : DLCO (expressed as absolute numbers and % predicted), kCO (expressed as absolute numbers and % predicted).

3.4.9. Patient reported outcomes (PROs): CAT® score (COPD Assessment Test), mMRC dyspnoea scale (modified Medical Research Council) 3.4.10. Imaging variables: a low-dose CT scan will be performed in each of the participants in the healthy smokers group and COPD, in order to determine the extent of the areas of emphysema (expressed as %LAA- percentage of Low-attenuation areas) and the airway compartment (expressed ad %WA- width of airway wall).

3.4.11. Blood biomarkers: a peripheral blood collection sample will be obtained in each participant in order to determine peripheral blood eosinophils (expressed as total eosinophil count & percentage from total leucocyte count), peripheral PMN (expressed as total PMN count & percentage from total leucocyte count), CPR (C- reactive protein) and fibrinogen.

3.4.12. CPCs isolation in peripheral blood: The CPCs isolation technique described above is actually protected by a provisional Spanish Patent Application (P201730724)

ELIGIBILITY:
Inclusion Criteria:

* Adults of >35 years-old.
* Patients who have given written informed consent
* Absence of respiratory infection or COPD exacerbation in the 4 previous weeks to baseline visit.

Exclusion Criteria:

* Other respiratory condition apart from COPD, such as previous diagnosis of bronchial asthma, obstructive sleep apnoea, idiopathic pulmonary fibrosis, pulmonary tuberculosis, alpha1 antitrypsin deficiency.
* Current or previous cancer history (even if the patient has been diagnosed >5 years and there is no evidence of recurrence of disease).
* Unwillingness to perform pulmonary function test or CT scan.
* Participation in another investigational study or clinical trial.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 healthy non-smokers, 30 healthy smokers and 100 patients with COPD (70 patients with mild to moderate disease- 35 of them below 60 years-old and 35 above 60 years-old-, and 30 patients with severe to very severe COPD -15 of them below 60 years-old and 15 above 60 years-old).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the prevalence of CPCs isolation in peripheral blood from COPD patients, smoking and non-smoking healthy controls with a patented liquid-biopsy technique. | 1 year

SECONDARY OUTCOMES:
Establish if there are differences between CPCs isolation rates from COPD patients, smoking and non-smoking healthy controls | 1 year
Evaluate the relationship between CPCs isolation and the degree of parenchymal destruction and empyshema expresed as DLCO and kCO | 1 year
Evaluate the relationship between CPCs isolation and emphysema degree expressed as CT scan measurements (% LAA). | 1 year
Evaluate the relationship between historical FEV1decline and CPCs isolation in COPD patients. | 2 year
Evaluate the relationship between prospective 1 year FEV1 decline and CPCs isolation in COPD patients. | 1 year
Evaluate the impact of CPCs isolation on deterioriation of HRQoL in COPD using CAT scores at baseline and change from baseline during 1 year follow- up. | 1 year

OTHER OUTCOMES:
Evaluate the rate of moderate and severe exacerbations during 1-year follow up between COPD patients with and without CPCs isolation after adjustment for confounding variables | 1 year
Evaluate the time to first moderate and severe exacerbation during 1-year follow up between COPD patients with and without CPCs isolation after adjustment for confounding variables. | 1 year
Evaluate if there are differences in the rate of CPCs isolation between those patients with early onset COPD (defined as those with COPD before 60 years of age) and those with normal onset COPD (defined as those with COPD after 60 years of age). | 1 year
Evaluate the impact of CPCs isolation on deterioriation of HRQoL in smoking subjects using CAT scores at baseline and change from baseline during 1 year follow- up. | 1 year
Evaluate the relationship between prospective 1 year FEV1 decline and CPCs isolation in smoking and non-smoking controls. | 1 year

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital de Alta Resolución de Loja, Loja, Granada
  - Hospital Universitario de Torrecardenas, Almería
  - Universidad de Granada- Facultad de Medicina, Granada
  - GENYO, centro Pfizer- Universidad de Granada- Junta de Andalucía de inestigación genómica y oncológica, Granada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: At the end of recruitment and analysis
Access Criteria: Upon reasonable request